CLINICAL TRIAL: NCT03567668
Title: Individualized Surgical Repair for Congenital Mitral Insufficiency in Infants and Children
Brief Title: Surgical Valvuloplasty for Congenital Mitral Insufficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hong Liu (Other)
Responsible Party: Sponsor-Investigator, Hong Liu, Clinical Investigator, Nanjing Medical University
Organization: Nanjing Medical University (Other)
Other Study IDs: TedaICH-MVP
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Mitral Insufficiency; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Mitral Valve Insufficiency; Pulmonary Arterial Hypertension | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mitral valvuloplasty — Commissural plication was the most commonly used technique to repair mitral insufficiency, which was selectively supplemented by a specific combination of one or more of the following procedures: cleft closure, chordal shortening, transposition or replacement, edge-to-edge repair, leaflet augmentation, or division of papillary muscles, depending on the individual etiology and anatomy.
  Other Names: mitral valve repair

SUMMARY:
Congenital mitral insufficiency is one of the most common valvular diseases in the pediatric population worldwide, carrying a high morbidity and mortality risk if not treated immediately and properly. Given that mitral replacement likely increased risk of cardiac dysfunction and mitral reoperation, mitral repair is the currently preferred surgical strategy in the majority of pediatric patients with mitral insufficiency. Unfortunately, previous evidences demonstrated the long-term hemodynamic alteration in response to significant mitral regurgitant might lead to a reversible or irreversible pulmonary vascular remodeling regardless of concomitant other cardiac malformations, which is associated with increased risk of morbidity and mortality following the surgery. Currently available researches mainly focused the association of pulmonary vascular pressures with risk of mortality and morbidity on adult rheumatic or degenerative mitral insufficiency; however, knowledge is still lacking regarding pediatric population with congenital mitral insufficiency. The investigator wil assess the relationship between baseline sPAP and risk of operative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* evidence of normal or preserved left ventricular systolic function (defined as left ventricular ejection fraction [LVEF] >50%);
* native mitral regurgitation of grade moderate or greater;
* with or without systemic-to-pulmonary shunting necessitating concomitant surgical repairs, regardless of pulmonary arterial pressure or pulmonary artery wedge pressure.

Exclusion Criteria:

* functional single ventricle;
* rheumatic mitral diseases;
* Eisenmenger syndrome;
* aortopathy, transposition of the great arteries, obstructions of ventricular outflow tract, malignant arrhythmias, cardiomyopathy, microbiological identification of infective endocarditis;
* a history of pericardiotomy or intervention therapy.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The infants and young children aged 5 months to 15 years are eligible for enrolment in this study if they had echocardiography confirmed mitral insufficiency.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival | Postoperatively; until five years after initial operation
  recurrence-free survival is defined as free of more than moderate mitral valve regurgitation

SECONDARY OUTCOMES:
Postoperative complications | Postoperatively, until one month after initial operation
  All postoperative complications and their treatment will be registered.

CONTACTS AND LOCATIONS:
Locations (1):
- TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalfa D, Vergnat M, Ly M, Stos B, Lambert V, Baruteau A, Belli E. A standardized repair-oriented strategy for mitral insufficiency in infants and children: midterm functional outcomes and predictors of adverse events. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1459-66. doi: 10.1016/j.jtcvs.2014.02.057. Epub 2014 Feb 26. PMID 24667029